CLINICAL TRIAL: NCT04734743
Title: Upper Extremity Muscle Strength and Endurance, Functional Capacity, Respiratory Function and Quality of Life in Child and Adolescent With Cystic Fibrosis
Brief Title: Muscle Strength, Functional Capacity, Respiratory Function and Quality Of Life In Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cagtay Maden (Other)
Responsible Party: Sponsor-Investigator, Cagtay Maden, Principal Investigator, physiotherapist, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016/06
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis; Muscle Strength; Pulmonary Function; Functional Capacity; Exercise Tolerance; Muscular Endurance
Keywords: muscle strength; pulmonary function; Cystic Fibrosis; functional capacity
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cystic fibrosis (Other)
  Interventions: Other: cystic fibrosis

INTERVENTIONS:
Other: cystic fibrosis — Evaluation of Upper Extremity Muscle Strength and Endurance, functional capacity, Respiratory Function and Quality of Life

SUMMARY:
This study was designed to investigate the relationship between upper extremity muscle strength and endurance, functional capacity, and quality of life child and adolescent with cystic fibrosis

DETAILED DESCRIPTION:
Child and adolescent with cystic fibrosis patients were assessed for upper extremity muscle strength and (Shoulder abductors muscle strength, Elbow flexion muscle strength, Handgrip strength) muscular endurance(arm pull-up test), lung function test, and functional capacity (six-minute walk test distance), and Quality Of Life (Cystic Fibrosis Questionnaire-Revised)

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with CF with clinical findings and gene mutations consistent with CF, having over 60mEq / L in two measurements in sweat chlorine examinations

Exclusion Criteria:

* Patients who did not exacerbate the disease in the last four weeks, who had good cooperation and did not have any orthopedic problems in the hand-shoulder-arm complex were included.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) | 1 day
  Pulmonary function tests were evaluated with a spirometer. It is the volume of air released in the first second from the beginning of the difficult vital capacity maneuver. In general, it gives information about the restriction in major airlines. FEV1 / FVC ratio decrease shows obstruction, FEV1 shows the severity of obstruction.
Six-minute walk test | 1 day
  In the 6-minute walk test (6MWT), subjects were asked to walk as fast as they could walk within 6 minutes along a 30-meter straight corridor. The test was performed twice within the same day at intervals of half an hour. The longer distance value for each patient from the two tests used was used for statistical analysis.
Forced Vital Capacity (FVC) | 1 day
  Pulmonary function tests were evaluated with a spirometer. It is the volume of air that comes out with rapid and powerful exhalation following deep inspiratory. Healthy people can normally extract 80 percent of their lung volume in 6 seconds or less
Peak Expiratory Flow (PEF) | 1 day
  Pulmonary function tests were evaluated with a spirometer. It is measured by the maximum exhalation maneuver following the maximum inspiration. It gives information about obstruction in large airways.
Upper Limb Muscle Strength | 1 day
  Evaluation of peripheral muscle strength Deltoideus (shoulder abduction), Biceps Brachii (elbow flexion) muscles were evaluated with a digital dynamometer (Lafeyette manual muscle tester, U.S.A). Handgrip strength was measured by a hand dynamometer (Baseline LITE hand dynamometer, U.S.A). In each muscle test, the right and left sides were evaluated separately and repeated three times and the best values obtained were recorded in Newton (N). Arithmetic means of the right and left sides were used for statistical analysis.
Upper Limb muscular endurance | 1 day
  The arm pull-up test was used in the evaluation of muscular endurance.
Ouality of Life | 1 day
  Cystic Fibrosis Questionnaire-Revised (CFQ-R) was used to evaluate the quality of life. There are four CFQ-R questionnaires for parents of children aged 6 years and over, three different age groups [6-10, 12-13, and over). The child's version of CFQ-R consists of 35 questions in 8 parts, Physical Functioning, Emotional Functioning, Social Functioning, Body Image, Eating Disturbances, Treatment Burden, Respiratory symptoms, and Digestive symptoms. Its values range from 0 to 100 points and the higher the score, the better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Çağtay maden, MSc, Pt, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu Universty, Gaziantep, Şahinbey, Turkey (Türkiye)